CLINICAL TRIAL: NCT05359900
Title: The Effect of Pain Education on Chiropractic Students' Understanding of Chronic Pain, Clinical Recommendations and Attitudes Towards People With Chronic Pain
Brief Title: The Effect of Pain Education on Chiropractic Students' Understanding of Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Collaborators: London South Bank University (Other); McTimoney College of Chiropractic (Unknown); AECC University College (Unknown); University of South Wales (Other)
Responsible Party: Principal Investigator, Paul Chesterton, Professor, Teesside University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TeessideUniversity22
Record Dates: First submitted 2022-03-11; First posted 2022-05-04 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Pain, Chronic; Education
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Multi-site, single-blind two arm, randomised control trial.
  The study would be conducted an five sites in total:
  Teesside University; The Welsh institute of Chiropractic - University of South Wales; The AECC University College; McTimoney College of Chiropractic; London Southbank University.
  Each site will follow the same protocol. Randomisation will occur at each individual site. Data will be pooled for analysis.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant information is pseudonymised using student numbers only. As soon is data is generated data will be fully anonymised.
  The outcome assessor will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain neuroscience education (Experimental): Pain neuroscience education group. One-off, 70 minute duration session delivered by Dr Cormac Ryan.
  Interventions: Other: Pain neuroscience education
- Red flag education (Active Comparator): Red flags education group. One-off 70 minute duration session delivered by Dr Cormac Ryan.
  Interventions: Other: Red Flag Education

INTERVENTIONS:
Other: Pain neuroscience education — Pain neuroscience education lecture
  Arms: Pain neuroscience education
Other: Red Flag Education — Red Flag education lecture
  Arms: Red flag education

SUMMARY:
Chronic pain is the leading cause of disability worldwide affecting just under 28 million people in the UK. Chronic pain conditions require a biopsychosocial rather than a biomedical model of care. Biomedical management lacks evidence of effectiveness but also has the potential to exacerbate the condition by raising fears and anxiety about potential pathological abnormalities.

Thus, the pre-registration phase is an important point where an individual's understanding of, and beliefs about, pain and people with pain may be shaped for the future. The need for improved and better education of healthcare professionals to support best practice for low back pain with the aim of integrating professionals' management of low back pain and fostering innovation in practice is well recognised. Pain education research with pre-registration chiropractors is lacking.

Therefore, this study aims to:

To compare the effect of two pain education intervention, through a multi-site randomised control trial, on the following three questionnaire based outcome measures:

1. Knowledge (understanding) of chronic pain
2. Attitudes towards chronic pain patients
3. Pain management behaviours

DETAILED DESCRIPTION:
In 2011 Briggs et al described pain education at undergraduate level for healthcare professionals as 'woefully inadequate'. Pain Neurophysiology Education (PNE) can improve undergraduates' pain understanding/management, however previous RCTs used single discipline groups and immediate follow-up. Investigation of the effectiveness of this education on students across the multi-professional team with medium-to-long-term follow-up will provide important new information on the generalisability of existing data and whether or not any changes in pain understanding/management are maintained over time.

This study aims to contribute to the development of neuromusculoskeletal chiropractic education by identifying whether or not this education, which aims to up skill healthcare professionals of the future, is effective and can change their behaviours in practice to enhance patient care in chronic pain management. PNE has been shown to be useful in patient care in conjunction with other treatment methods. If this intervention is successful in altering pain attitudes and knowledge in keeping with modern science then students may feel more confident and able to manage pain post qualification. The findings of this study will support or refute the addition of PNE into healthcare professional undergraduate programmes

ELIGIBILITY:
Inclusion Criteria:

* Current Chiropractic students enrolled at either: Teesside University; The Welsh institute of Chiropractic - University of South Wales; The AECC University College; McTimoney College of Chiropractic; London Southbank University
* Willing to consent to attending two educational sessions followed by completing questionnaires

Exclusion Criteria:

* Chiropractic students not actively enrolled at either: Teesside University; The Welsh institute of Chiropractic - University of South Wales; The AECC University College; McTimoney College of Chiropractic; London Southbank University
* Participants will be excluded if they have previously received in depth education on red flags and or pain neurophysiology.
* Students not willing to consent to attending two educational sessions followed by the completion of questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
The 12-item Revised Pain Neurophysiology Quiz (change assessed) | Immediate and 6-month follow-up
  This is a validated tool for assessing knowledge of pain physiology. Measures knowledge of pain physiology using a 12 point validated questionnaire. Low score is poor sign. Scores range from 0-12.
The 10-item Red Flags knowledge questionnaire (change assessed) | Immediate and 6-month follow-up
  This is a questionnaire containing 10 yes/no questions to assess participants knowledge of red flags. Low score is a poor sign. Scores range from 0-10.
The 13-item Health Care Providers' Pain and Impairment Relationship Scale (HC-PAIRS) (change assessed) | Immediate and 6-month follow-up
  this a validated measure of health care professionals attitudes towards the ability of patients with pain to function despite their pain. The Health Care Providers Pain and Impairment Relationship Scale assesses attitudes and beliefs towards pain using a 13 item validated questionnaire. High score is a worse outcome. Scores range from 13-91.
Case vignette (change assessed) | Immediate and 6-month follow-up
  Measures clinical practise behaviours in pain management. A validated proxy measure of clinical behaviour, MCQ weighted as appropriate or inappropriate according to current national clinical guidelines. A low score is considered good, and scores range from 4 to 20.

SECONDARY OUTCOMES:
Semi-structured Interviews | 6-month follow-up
  Participants will be invited to take part in a semi-structured interview based in realtion to their knowledge retention and subject understanding.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - McTimoney College of Chiropractic, Abingdon
  - The AECC University College, Bournemouth
  - London Southbank University, London
  - The Welsh institute of Chiropractic - University of South Wales, Pontypridd

IPD SHARING:
Plan to Share IPD: No